CLINICAL TRIAL: NCT07270679
Title: Genetic Markers of Susceptibility to Chemotherapy-induced Ovarian Damage in Cancer Patients Undergoing Ovarian Biopsy for Cryopreservation.
Status: Recruiting | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Sponsor
Other Study IDs: GTM_OCP; FERR24RD (Other Grant/Funding Number: Ferring S.p.A.)
Record Dates: First submitted 2025-11-26; First posted 2025-12-08 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-07

CONDITIONS: Breast Cancer; Hodgkin Lymphoma
MeSH Terms: conditions — Breast Neoplasms; Hodgkin Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Ovarian tissue stored in the cryobank from oncology patients who underwent fertility preservation through ovarian tissue cryopreservation prior to undergoing gonadotoxic therapies. The portion of the biological material designated for reproductive or hormonal purposes will not be used; instead, a part of the ovarian tissue sample already allocated by institutional procedure for laboratory analyses will be utilized.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Italian Cancer Registry data show a steady increase in the number of cancer survivors due to advances in treatment. However, these treatments can impair ovarian function, causing premature ovarian insufficiency (POI). Women with POI may experience vasomotor symptoms, infertility, psychological distress, and a significant reduction in quality of life. POI typically occurs before age 40 and is characterized by irregular menstruation and biochemical alterations (elevated gonadotropins and low estradiol). Chronic estrogen deficiency in POI is associated with increased risks of cardiovascular disease, cognitive decline, osteoporosis, psychological issues, and reproductive dysfunction.

Preliminary studies suggest that chemotherapy-induced POI results from genetic changes in ovarian tissue, indicating a crucial role of genetic variations in individual susceptibility. Incidence rates of POI vary widely: about 38% after Hodgkin lymphoma and between 15% and 94% after breast cancer. Currently, there is no personalized pre-treatment risk assessment, complicating informed decision-making regarding ovarian function and fertility.

Fertility preservation options include ovarian tissue and oocyte cryopreservation. This study aims to compare the mutational status of DNA repair genes in ovarian tissue fragments from women who underwent ovarian cryopreservation and completed chemotherapy for lymphoma or breast cancer, categorized into those who developed POI and those who did not. Additionally, the mutational load of these genes will be compared between groups.

The study includes patients aged 18-38 who preserved ovarian tissue before gonadotoxic therapy between 2002 and 2024 at the IRCCS Azienda Ospedaliero-Universitaria di Bologna, Policlinico di S. Orsola. Two groups will be analyzed:

Group 1: Patients who developed POI after gonadotoxic treatment

Group 2: Patients who did not develop POI

Group assignment will be based on clinical and anamnesis data. Cryopreserved ovarian tissue from all participants will undergo advanced molecular analyses by Next Generation Sequencing (NGS) to assess germline and somatic mutational status and load. The genetic variant analysis, conducted in collaboration with the Computational Genomics Unit of IRCCS AOUBO, will focus on a panel of 26 DNA repair genes. Bioinformatic analysis will be performed using the Ion Reporter platform, with clinically relevant variants validated by orthogonal methods.

The study plans to enroll approximately 50 patients, 25 per group.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 and ≤ 38 years at the time of cryopreservation
* Patient diagnosed with breast cancer or lymphoma, who underwent ovarian biopsy and cryopreservation of ovarian tissue prior to the initiation of gonadotoxic treatment
* Gonadotoxic therapy completed at least 6 months prior
* Written informed consent obtained for participation in the study and for the processing of personal, sensitive, and genetic data

Exclusion Criteria:

* Patients with a history of gonadotoxic treatments prior to ovarian tissue cryopreservation
* Patients undergoing hormonal therapy that suppresses ovarian function (e.g., GnRH analogs)
* Presence of other conditions potentially responsible for premature ovarian insufficiency [e.g., BRCA1 and BRCA2 mutations, Li-Fraumeni syndrome, Bloom syndrome, Fanconi anemia, Fragile X syndrome, Cowden syndrome, Lynch syndrome (Hereditary Non-Polyposis Colorectal Cancer - HNPCC), Ataxia-Telangiectasia]
* Family history of premature ovarian insufficiency

Ages: 18 Years to 38 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Reproductive-age patients undergoing chemotherapy treatment for breast cancer or lymphoma, following ovarian biopsy and ovarian tissue cryopreservation at the Cryobank Laboratory for Ovarian Tissue Cryopreservation and Cell Cultures of the Unit of Gynecology and Human Reproductive Pathophysiology, IRCCS Azienda Ospedaliero-Universitaria di Bologna, Policlinico di S. Orsola
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-07-23 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-12-03 (Estimated)

PRIMARY OUTCOMES:
To compare the mutational status of genes involved in DNA repair mechanisms in ovarian tissue fragments from women who underwent ovarian cryopreservation and completed chemotherapy treatment for lymphoma or breast cancer | At least 6 months after the end of chemotherapy
  Onset of POI (Premature Ovarian Insufficiency)

SECONDARY OUTCOMES:
To compare the mutational load of altered genes between women who developed POI and those who did not after undergoing chemotherapy | At least 6 months after the end of chemotherapy
  Onset of POI

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Azienda Ospedaliero-Universitaria di Bologna, Bologna, Bologna, Italy

IPD SHARING:
Plan to Share IPD: No